CLINICAL TRIAL: NCT04555304
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Phase 2 Study of Weekly Paclitaxel With or Without KH903 in Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma, Refractory to or Progressive After First-Line Therapy With Platinum and Fluoropyrimidine
Brief Title: Phase 2 Study of KH903 in Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma As Second-Line Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KH903-40101-CRP
Record Dates: First submitted 2020-08-05; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Gastric Cancer; Gastroesophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — KH902 fusion protein; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KH903 + Paclitaxel (Experimental): IV KH903 4 mg/kg IV paclitaxel 80 mg/m²
  Interventions: Drug: KH903 + Paclitaxel
- Placebo + Paclitaxel (Active Comparator): IV Placebo IV paclitaxel 80 mg/m²
  Interventions: Drug: Placebo + Paclitaxel

INTERVENTIONS:
Drug: KH903 + Paclitaxel — KH903 4 mg/kg will be administered intravenously on D1 D8 D15and D22 in a 28-day cycle； Paclitaxel 80 mg/m² will be administered intravenously on D1, D8 and D15 in a 28-day cycle
  Arms: KH903 + Paclitaxel
Drug: Placebo + Paclitaxel — Placebo will be administered intravenously on D1 D8 D15and D22 in a 28-day cycle； Paclitaxel 80 mg/m² will be administered intravenously on D1, D8 and D15 in a 28-day cycle
  Arms: Placebo + Paclitaxel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the study drug known as KH903 in participants with gastric and gastroesophageal cance

ELIGIBILITY:
Inclusion Criteria:

* 1.Prior to any detailed procedures of this study, subjects are able to understand, voluntarily participate in and sign the informed consent approved by the ethics committee.
* 2.Age ≥ 18 years.
* 3.Histologically confirmed, unresectable, locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma .
* 4.Have at least 1 measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.
* 5.Have experienced documented objective radiographic or symptomatic disease progression during first-line therapy, or within 4 months after the last dose of first-line therapy with any platinum or/and fluoropyrimidine doublet for unresectable or metastatic disease.Second line chemotherapy is suitable for paclitaxel.
* 6.Laboratory test values must meet the following criteria. ANC ≥1.5×109/L, platelets ≥ 100×109/L, hemoglobin≥9g/dL. Blood creatinine ≤ 1.5 ×ULN or creatinine clearance ≥ 50 mL/min/m2. Total bilirubin ≤ 1.5× ULN(≤ 3 x ULN if Gilbert disease), AST and ALT ≤ 2.5× ULN (≤ 5×ULN if hepatic metastasis).

INR ≤ 1.5× ULN, APTT ≤ 1.5× ULN. Dipstick proteinuria <2+ or 24 hour proteinuria <1g .

* 7.Good performance status Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 to 1.
* 8.Life expectancy of ≥ 3 months.

Exclusion Criteria:

* 1.Histologically confirmed squamous cell carcinoma or undifferentiated gastric cancer.
* 2.Patients with disease progression within 6 months after previous adjuvant or neoadjuvant chemotherapy with paclitaxel, or patients with recurrent or metastatic gastric adenocarcinoma or GEJ adenocarcinoma treated with paclitaxel.
* 3. GI perforation and/or fistulae in the 6 months preceding randomization.
* 4.Deep-vein thrombosis, pulmonary embolism (PE), or any other episode of Uncontrolled thromboembolism in the 6 months preceding randomization.
* 5.Any arterial thromboembolic event (such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack)
* 6.Uncontrolled hypertension (≥150/100 mm Hg ) despite properly observed antihypertensive therapy.
* 7.Known brain metastasis.
* 8.Known allergy to paclitaxel or KH903.
* 9.Serious concurrent infection or medical illness.
* 10.Active hepatitis B virus or Active hepatitis C virus (HCV) infection at screening.
* 11.Any condition which results in an undue risk for the patient during the trial participation according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | Time from date of randomization until the date of first documented Progression or date of death from any cause， whichever came frist，assessed up to18 months
  Date of randomization until the date of first documented Progression or date of death from any cause， whichever came first

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from date of randomization until the date of first documented CR or PR，assessed up to18 months
  Percentage of Participants with a Best Overall Response (BOR) of Partial Response (PR) or Complete Response (CR)
Duration of Response (DOR) | Time from first documented evidence of CR or PR until the date of first documented progression ，assessed up to18 months
  is defined as the time from first documented evidence of CR or PR until the date of first documented progression as assessed by RECIST 1.1 or death; assessed up to18 months
Disease Control Rate (DCR) | Time from date of randomization until the date of first documented Progression，assessed up to18 months
  Percentage of Participants who have achieved CR, PR and SD to study treatment;
AE | AEs（NCI CTCAE 5.0） collected at each cycle，Assessed up to18 months
  Number of Subjects with treatment-related adverse events (AEs)Defined by all

CONTACTS AND LOCATIONS:
Overall Officials: yi ba, PhD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital